CLINICAL TRIAL: NCT05035407
Title: A Phase I Trial of T Cell Receptor Gene Therapy Targeting KK-LC-1 for Gastric, Breast, Cervical, Lung and Other KK-LC-1 Positive Epithelial Cancers
Brief Title: T Cell Receptor Gene Therapy Targeting KK-LC-1 for Gastric, Breast, Cervical, Lung and Other KK-LC-1 Positive Epithelial Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Site plans to become a site for a multicenter study of this therapy
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000045; 000045-C
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Kita-kyushu Lung Cancer Antigen 1, Human
Keywords: Vaccine; Gene Therapy; Cell Therapy; T Cell Therapy; Immunotherapy; CAR T; Tumor infiltrating lymphocyte; Triple Negative Breast Cancer; Metastatic Solid Tumor; Metastatic carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis; Carcinoma | interventions — Interleukin-2; aldesleukin; Cyclophosphamide; fludarabine; fludarabine phosphate; Electrocardiography; Diagnostic Imaging; Tomography, X-Ray Computed; Magnetic Resonance Imaging; Positron-Emission Tomography; Biopsy; Acetaminophen; Ondansetron; Meperidine; Indomethacin; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment at Dose Levels 1 through 6 (Experimental): Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  Interventions: Drug: IL-2 (Aldesleukin); Drug: Cyclophosphamide; Biological: KK-LC-1 TCR; Drug: Fludarabine; Diagnostic Test: EKG; Diagnostic Test: CXR; Diagnostic Test: CT; Diagnostic Test: MRI; Diagnostic Test: PET; Procedure: Biopsy; Drug: Acetaminophen; Drug: Ondansetron; Drug: Meperidine; Drug: Indomethacin; Drug: Famotidine

INTERVENTIONS:
Drug: IL-2 (Aldesleukin) — Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Other Names: Interleukin-2 (Aldesleukin)
Drug: Cyclophosphamide — 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  Other Names: Cytoxan
Biological: KK-LC-1 TCR — Transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells in escalating doses.
  Dose Level 1: 1 x 10^8 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Dose Level 2: 5 x 10^8 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Dose Level 3: 1 x 10^9 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Dose Level 4: 5 x 10^9 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Dose Level 5: 1 x 10^10 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Dose Level 6: 6 x 10^10 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Other Names: Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor
Drug: Fludarabine — 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  Other Names: Fludara
Diagnostic Test: EKG — At screening/baseline.
  Other Names: Electrocardiogram
Diagnostic Test: CXR — At screening/baseline.
  Other Names: Chest x-ray
Diagnostic Test: CT — At screening/baseline.
  Other Names: Computed tomography
Diagnostic Test: MRI — At screening/baseline
  Other Names: Magnetic resonance imaging
Diagnostic Test: PET — At screening/baseline.
  Other Names: Positron emission tomography
Procedure: Biopsy — Optional. At screening/baseline. And (+/- 48 hours) prior to start of chemo, at the first response assessment visit and at time of progression.
  Other Names: Bx
Drug: Acetaminophen — 650mg every(q) 4 hours for supportive therapy as needed.
  Other Names: Tylenol; Panadol
Drug: Ondansetron — 0.15mg/kg/dose intravenous every(q) 8 hours for nausea and vomiting.
  Other Names: Zofran; Zofran ODT; Zuplenz
Drug: Meperidine — 25-50mg intravenous for severe chilling if needed.
  Other Names: Demerol
Drug: Indomethacin — 50-75mg every(q) 8 hours for supportive therapy as needed.
  Other Names: Tivorbex; Indocin
Drug: Famotidine — 20mg every(q) 12 hours for supportive therapy as needed.
  Other Names: Pepcid; Acid reducer; Acid controller

SUMMARY:
Background:

Researchers have found a new way to treat cancer using T cell therapy. The therapy used in this study is T Cell Receptor (TCR) Gene Therapy Targeting Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1), a cancer germline antigen that is expressed by certain cancers. This therapy is a type of treatment in which participants T cells (a type of immune system white blood cell) are changed in the laboratory to attack cancer cells and given back to the participant. This treatment might help people with KK-LC-1 positive cancers which may include gastric, breast, cervical, lung and other epithelial Cancers. Epithelial cancers are cancers that begin in the cells that line an organ.

Objective:

The purpose of this study is to determine the safety of different doses of KK-LC-1 TCR T cells plus aldesleukin to treat metastatic or refractory/recurrent KK-LC-1 positive cancers.

Eligibility:

Adults aged 18 and older with metastatic or refractory/recurrent KK-LC-1 positive epithelial cancer.

Design:

Participants will be screened with human leukocyte antigen (HL)typing (a blood test needed for eligibility) and KK-LC-1 testing of the cancer tumor (to determine if the cancer is KK-LC-1 positive). A new biopsy may be needed if tumor from an outside location is not available for KK-LC-1 testing. Eligible participants will come to the National Institutes of Health (NIH) campus to have a screening evaluation which will include physical exam, review of medical history and current medications, blood and heart tests, imaging (X-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI) or positron emission tomography (PET) scan), and evaluation of participants veins that are used for drawing blood.

If the participant is eligible for the study based on the screening evaluation, they will have a baseline evaluation prior to receiving the experimental treatment which may include additional laboratory or imaging tests.

Participants will have a large intravenous (IV) catheter inserted into a vein to undergo a procedure called leukapheresis. Leukapheresis is the removal of the blood by a machine to collect specific white blood cells. The remaining blood is returned to the body. This procedure is needed to collect the cells that will be modified to target the cancer. The cells are grown in the lab and given back to the participant through an injection into the participant's tumor. It takes 11-15 days to grow the cells.

While the cells are growing, the participant will be admitted to the hospital about one week

before the cell infusion to receive 2 types of chemotherapy through an IV catheter over 5 days. The main purpose of the chemotherapy is to make the cells more effective in fighting the cancer tumors. The cells will be given 1-2 days after the last dose of chemotherapy. Within 24 hours after the cell infusion, participants will be given a cell growth factor called aldesleukin through an IV for up to 4 days. Aldesleukin is thought to help the cells live longer in the participant's body. Participants will recover in the hospital until they are well enough to go home, which is usually about 7-12 days after the cell infusion or last dose of aldesleukin.

Participants will have a follow-up visit at approximately 40 days after the date of cell infusion. This visit will be to evaluate the safety of the cell therapy and the response of the cancer to the treatment which will include physical examination, lab tests, and imaging studies. If a participant has stable disease or their cancer has responded to the treatment, they will be seen again at 12 weeks post cell infusion, every 3 months x 3 visits, and then every 6 months x 5 years. If a participants cancer progresses after this therapy, they will be return to their home doctor for further management.

After receiving cell therapy, participants will be followed on a long-term gene therapy protocol. Participants will have blood drawn periodically to test if the cells have grown or changed. These blood tests will take place immediately before the cells, and then at 3, 6, and 12 months for the first year and possibly annually thereafter based on the results. These tests can be drawn locally and sent to the NIH. After a participant is off the study, they will be contacted by telephone or mailed questionnaire for a total of 15 years after cell therapy....

DETAILED DESCRIPTION:
Background:

Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) is a cancer germline (CG) antigen with expression restricted to germ cells (which lack major histocompatibility complex (MHC) class I expression) in adults and epithelial cancers including lung, breast and gastric.

This limited expression pattern makes it an ideal target for T Cell Receptor (TCR) gene therapy.

TCR T cell therapy targeting CG antigens has been shown to induce objective responses without autoimmunity or off-target toxicity in participants with melanoma, synovial sarcoma and cervical cancer.

T cells genetically engineered with a TCR targeting KK-LC-1 display specific reactivity against HLA-A01:01 (human leukocyte antigen serotype within HLA-A "A" serotype group), KK-LC-1 target cells.

KK-LC-1 TCR T cells can mediate tumor regression in pre-clinical mouse models of cancer.

Objective:

To determine the maximally tolerated dose of KK-LC-1 TCR T cells plus aldesleukin for the treatment of metastatic KK-LC-1 positive epithelial cancers.

Eligibility:

Participants greater than or equal to 18 years old with metastatic or refractory/recurrent KK-LC-1 positive epithelial cancer.

Prior first line systemic therapy is required unless the participant declines standard treatment.

Participants must be HLA-A-01:01-positive.

Design:

This is a phase I clinical trial that will test the safety and efficacy of escalating doses of KK-LC-1 TCR T cells.

Participants will receive a non-myeloablative lymphocyte-depleting preparative regimen of cyclophosphamide and fludarabine followed by a single infusion of KK-LC-1 TCR T cells and high-dose aldesleukin.

Re-treatment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) positive epithelial cancer (KK-LC-1 positivity assay performed at Rutgers Cancer Institute of New Jersey). KK-LC-1 expression will be determined by immunohistochemistry (IHC). KK-LC- 1 score of 25% or greater will be considered positive.
* Participants must be HLA-A 01 (human leukocyte antigen serotype within HLA-A "A" serotype group) by low resolution typing, and HLA-A 01:01 by one of the high-resolution type results
* Measurable metastatic or refractory/recurrent KK-LC-1+ epithelial cancer (determined by Immunohistochemistry (IHC).
* All participants must have received prior first line standard therapy or be ineligible to receive available therapies with known survival benefit.
* Participants with three or fewer brain metastases that have been treated with surgery or stereotactic radiosurgery are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month before protocol treatment. Participants with surgically resected brain metastases are eligible.
* Age >18 years of age. Because no dosing or adverse event data are currently available on the use of KK-LC-1 T cell receptor (TCR) in participants <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status <1.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL
  * platelets >=100,000/mcL
  * hemoglobin >=9.0 g/dL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) =<2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits

OR

* creatinine clearance >=60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.

  -Serology:
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the participant must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.

  * The effects of the study agent on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, individuals of child-bearing potential and their partners must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and up to twelve (12) months after treatment. Individuals of childbearing potential must have a negative pregnancy test. Individuals of childbearing potential are defined as all individuals except individuals who are postmenopausal or who have had a hysterectomy. Postmenopausal will be defined as individuals over the age of 55 who have not had a menstrual period in at least one year or a participant that has received a treatment (i.e., chemotherapy or pelvic radiation) that has resulted in them becoming postmenopausal. Should an individual become pregnant or suspect pregnancy while individuals or partner is participating in this study, individuals should inform treating physician immediately.
  * Because there is a potential risk for adverse events in nursing infant's secondary to treatment of the mother with KK-LC-1 TCR transduced peripheral blood lymphocytes (PBLs), breastfeeding should be discontinued if the mother is treated with KK-LC-1 TCR transduced PBL. These potential risks may also apply to other agents used in this study.
  * More than four weeks must have elapsed since any prior systemic therapy at the time the participant receives the KK-LC-1 TCR T cells.
  * Participants may have undergone minor surgical procedures within the past three weeks, as long as all toxicities have recovered to Grade 1 or less
  * Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents.
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine or aldesleukin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Participants with abnormal pulmonary function tests but stable obstructive or restrictive pulmonary disease may be eligible.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Participants with autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis or pancreatitis, and systemic lupus rythematosus. Hypothyroidism, vitiligo and other minor autoimmune disorders are not exclusionary.
* Participants on active systemic immunosuppressive therapy that cannot be safely withheld.
* Participants with a history of coronary revascularization or ischemic symptoms unless participant has a normal cardiac stress test.
* Any condition which would, in the opinion of the Principal Investigator, indicate that the subject is a poor candidate for the clinical trial or would jeopardize the subject or the integrity of the data obtained.
* Documented left ventricular ejection fraction (LVEF) <= 45%

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000045-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 1 x 10^8 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
- 5 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 5 x 10^8 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  No participants were enrolled at this dose level.
- 1 x 10^9 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 1 x 10^9 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  No participants were enrolled at this dose level.
- 5 x 10^9 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 5 x 10^9 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  No participants were enrolled at this dose level.
- 1 x 10^10 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 1 x 10^10 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  No participants were enrolled at this dose level.
- 6 x 10^10 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells: Non-myeloablative, lymphocyte depleting preparative regimen, followed by Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptors (TCRs) T cells plus aldesleukin at escalating doses
  IL-2 (Aldesleukin): Dose of 720,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period beginning within 24 hours of cell infusion and continuing for up to four days (maximum 12 doses).
  Cyclophosphamide: 30 mg/kg intravenous (IV) infusion over 1 hour (+ 10 min) Once daily x 2 doses (Days -6 and -5)
  KK-LC-1 TCR: 6 x 10^10 transduced Kita-Kyushu Lung Cancer Antigen-1 T-Cell Receptor (KK-LC-1) (TCR) T cells.
  Fludarabine: 25 mg/m^2 intravenous (IV) infusion over 30 minutes (+ 10 min) to be administered following completion of cyclophosphamide. Once daily x 5 doses (Days -6, -5, -4, -3, -2).
  No participants were enrolled at this dose level.
Period: Overall Study
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells | 5 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells | 1 x 10^9 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells | 5 x 10^9 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells | 1 x 10^10 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells | 6 x 10^10 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells
Started | 36 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 36 | 0 | 0 | 0 | 0 | 0
Not completed — Consented/enrolled on screening only. No participants signed the treatment consent for this study | 36 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.81 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 18
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) of Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T Cell Receptor (TCR) T Cells Plus Aldesleukin for the Treatment of KK-LC-1 Plus Cancers
Description: The MTD is the highest dose at which < 1 of 6 participants experienced a DLT or the highest dose level studied if 2 DLTs are not observed at any of the dose levels. A DLT is all grade 3 and greater toxicities related to cell infusion, with the exception of: Cytokine Release Syndrome (CRS) that resolves < grade 2 within 14 days of the last dose of aldesleukin; Autoimmune toxicity that resolves < grade 2 within 14 days from starting symptoms treatment (e.g. steroids); Cardiac, gastrointestinal, dermatological, hepatic, pulmonary, renal, hematologic, neurologic toxicity, or toxicity specified in the protocol attributable to aldesleukin that resolves to grade 2 within 14 days of the last dose of aldesleukin; and Transient grade 3 hypoxia associated with cell infusion that corrects to < grade 2 with supplemental oxygen and/or that resolves to < grade 2 within 24 hours; and Hemorrhage due to underlying cancer or prior radiotherapy.
Time Frame: 3 months
Population: No participants were treated, so MTD was not determined.
Measure: Number; unit: cells
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells
Number analyzed (Participants) | 0

2. Primary Outcome: Proportion of Participants Who Experience a Dose Limiting Toxicity (DLT) With the Number and Grade of Each Type of DLT
Description: A DLT is all grade 3 and greater toxicities related to cell infusion, with the exception of: Cytokine Release Syndrome (CRS) that resolves < grade 2 within 14 days of the last dose of aldesleukin; Autoimmune toxicity that resolves < grade 2 within 14 days from starting symptoms treatment (e.g. steroids); Cardiac, gastrointestinal, dermatological, hepatic, pulmonary, renal, hematologic, neurologic toxicity, or toxicity specified in the protocol attributable to aldesleukin that resolves to grade 2 within 14 days of the last dose of aldesleukin; and Transient grade 3 hypoxia associated with cell infusion that corrects to < grade 2 with supplemental oxygen and/or that resolves to < grade 2 within 24 hours; and Hemorrhage due to underlying cancer or prior radiotherapy. Toxicities were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: At the time of cell infusion, up to 30 days after cell infusion
Population: No participants were treated.
Measure: Number; unit: proportion of participants
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events (AEs) will be documented from the start date of chemotherapy through 40 days after the cell administration. Beyond 40days after the cells were administered, only AEs which are serious & related to the study intervention need to be recorded.
Population: The definition of an adverse event (AE) is "any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product…". Since participants on screening aren't administered a drug, then the definition of AE does not apply to them (per the protocol).
Measure: Count of Participants; unit: Participants
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 1 month. Since no participants were treated, per protocol, no data was collected on adverse events. Adverse events will be documented from the start date of chemotherapy through 40 days after the cell administration. Beyond 40 days after the cells were administered, only adverse events which are serious and related to the study intervention need to be recorded.
Description: The definition of an adverse event (AE) is "any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product…". Since participants on screening aren't administered a drug, then the definition of AE does not apply to them (per the protocol).
Arm/Group | 1 x 10^8 Transduced Kita-Kyushu Lung Cancer Antigen-1 (KK-LC-1) T cell receptor (TCR) T cells
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT05035407/Prot_SAP_000.pdf
  • Informed Consent Form: Treatment Affected Patient (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05035407/ICF_001.pdf
  • Informed Consent Form: Screening Consent (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05035407/ICF_002.pdf